CLINICAL TRIAL: NCT00826800
Title: A Pilot Study of Neoadjuvant FOLFOX Plus Bevacizumab Chemotherapy in Patients With Locally Advanced Colon Cancer
Brief Title: Neoadjuvant FOLFOX Plus Bevacizumab Chemotherapy in Patients With Locally Advanced Colon Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-162
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Colon Cancer
Keywords: BEVACIZUMAB (AVASTIN); FLUOROURACIL; LEUCOVORIN; OXALIPLATIN; Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Folfox protocol; Bevacizumab

ARMS (1):
- Neoadjuvant FOLFOX Plus Bevacizumab (Experimental): FOLFOX and bevacizumab will be given to colon cancer patients for 4 cycles over 8 weeks; an additional 2 cycles of FOLFOX without bevacizumab will be given for a total of 12 weeks of pre-operative chemotherapy.Restaging will be performed within 3 weeks of the 6th chemotherapy cycle. Colon surgery will be performed between weeks 3 and 6 subsequent to the 6th cycle of FOLFOX. Patients receiving preoperative chemotherapy without radiation will wait a minimum of 3 weeks from their last dose of chemotherapy, and 6 weeks from their last dose of bevacizumab, before proceeding to surgery. Specifically, it is intended that patients will undergo surgery between 3-6 weeks from completion of their neoadjuvant therapy as deemed clinically appropriate by their surgeon and medical oncologist. This permits a 7-10 week interval between the 4th bevacizumab administration and colon surgery.
  Interventions: Drug: FOLFOX and bevacizumab

INTERVENTIONS:
Drug: FOLFOX and bevacizumab — The patient will receive six treatments, two weeks apart. On each treatment day you will get Oxaliplatin, 5-FU,Leucovorin. On the first four treatments you will also get Bevacizumab (Avastin). These drugs are given through a Mediport. They will be given in an outpatient chemotherapy unit. Each tx will take about 4 hours. A pump for the 5-FU is worn around your waist. This drug is given over 2 days. Part II: Colon Cancer Surgery is standard practice, and is not a research procedure.Part III: Post-operative Re-Evaluation and Recovery The doctor will decide on the type of chemotherapy based on how the patient responded to the first chemotherapy. The plan will be for the patient to get 6 more doses of FOLFOX, without any further bevacizumab, unless your doctor finds a reason to do otherwise.

SUMMARY:
The purpose of this study is to see if giving chemo-therapy for colon cancer before surgery can shrink the cancer and lead to a higher rate of cure than operating first and then giving chemotherapy. Standard treatment for colon cancer is to first operate, and then, if the tumor is advanced, give chemotherapy for about 6 months. However, surgery delays the time until chemotherapy can start, since the body needs time to heal from the operation. During this time any cancer cells that remain in the body that were not removed by the operation may be allowed to grow. Giving chemotherapy first could attack the cancer cells right from the start, not only at the tumor site that we know of, but also at the site of any cancer cells that may have spread to other parts of the body. Another possible reason why giving chemo therapy first might work better is that the blood vessels that feed the cancer cells are intact before surgery and thus chemotherapy can travel directly to the cancer.

This study will also use the drug bevacizumab, in addition to the standard chemotherapy. Bevacizumab has been on the market since 2004 for colon cancer that has spread to other organs, but its use in earlier stage colon cancer, as planned in this trial, is still under study.

ELIGIBILITY:
Inclusion Criteria:

* NOTE: Patients may sign consent and be registered for this protocol prior to completion of assessment of criteria 6.1.1 and 6.1.2, (assuming all other eligibility criteria are met) so that endocolonic ultrasound and biopsy may be performed on study; as these procedures may be necessary to determine TNM staging and/or histopathology; however criteria 6.1.1 and 6.1.2 must be successfully met prior to patient receiving chemotherapy on this trial.
* 6.1.1 Clinical T1N1-2/T2N1-2/T3N0/T3N1-2/T4Ni-N2 adenocarcinomas of the colon determined by endocolonic ultrasound (ECUS) performed at MSKCC.
* 6.1.2 Colonoscopy with endoscopic biopsy of tumor at MSKCC for disease confirmation and correlative studies. Pathological confirmation of adenocarcinoma or poorly differentiated carcinoma as the primary histology.
* CT or MRI scans (done within 30 days of registration) of the Chest, Abdomen and Pelvis all without clear evidence of distant metastatic (M1) disease.
* Candidates for systemic therapy with FOLFOX and bevacizumab based on the opinion of the primary treating medical oncologist.
* Candidates for complete surgical resection prior to administration of any therapy.
* Performance status of ECOG 0 or 1.
* Patients must be of age ≥18 years.
* ANC ≥ 1.5 cells/mm3, PLT >150,000/mm3.
* Serum creatinine < or = to 1.5 OR creatinine clearance (measured or calculated) greater than 60 ml/min.

Exclusion Criteria:

* Primary tumor clearly unresectable.
* Tumors with neuroendocrine histology.
* Patients with tumors that require placement of an endocolonic stent prior to treatment initiation.
* Patients with a history of stroke or TIA.
* Patients with history of thrombotic episodes such as deep venous thrombosis, pulmonary embolus, MI, or CVA occurring more than 12 months prior to enrollment may be considered for protocol participation provided that they are on stable doses of anticoagulant therapy. Similarly, patients anticoagulated for atrial fibrillation or other conditions may participate provided that they are on stable dose of anticoagulant therapy. Clinicians must note the higher risk of bevacizumab therapy amongst patients with history of thromboembolic disorders and consideration for participation is at the discretion of the treating physician.
* No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matrix metalloprotease inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibody or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
* Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 6 months after the study. Subjects who are men must also agree to use effective contraception.
* Note: Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 6 months after the study in such a manner that the risk of pregnancy is minimized.
* WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35mIU/mL]. Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.
* Women who are pregnant or breast feeding. Note: women with a positive pregnancy test on enrollment or prior to study drug administration will be removed from study.
* Patients with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make the patient inappropriate for entry into this study.
* Patients with a history in the past five years of a prior malignancy, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Inadequately controlled, persistent (on more than one occasion) hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg).
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture (adjuvant trials: bone fractures must be healed
* Proteinuria as demonstrated by a UPC ratio ≥ 1.0 at screening
* Known hypersensitivity to any component of bevacizumab

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saltz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 01/19/2009 Protocol Closed to Accrual: 04/13/2010 Primary Completion Date (if applicable): 12/28/2010 Recruitment Location is the medical clinic
Groups:
- Neoadjuvant FOLFOX Plus Bevacizumab: FOLFOX and bevacizumab: The patient will receive six treatments, two weeks apart. On each treatment day patient will get Oxaliplatin, 5-FU,Leucovorin. On the first four treatments, patient will also get Bevacizumab (Avastin).
Period: Overall Study
Arm/Group | Neoadjuvant FOLFOX Plus Bevacizumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant FOLFOX Plus Bevacizumab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Pathologic Complete Response (Path CR) Rate in Patients With Locally Advanced (Stage II or III) Colon Cancer to FOLFOX-bevacizumab Administered as Neoadjuvant.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Neoadjuvant FOLFOX Plus Bevacizumab
Number analyzed (Participants) | 2
participants
  Complete Response | 1
  Partial Response | 1

ADVERSE EVENTS:
Arm/Group | Neoadjuvant FOLFOX Plus Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant FOLFOX Plus Bevacizumab (N=2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4)
Alkaline phosphatase increased (Investigations) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (13)
Anemia (Blood and lymphatic system disorders) | 2 (19)
White blood cell decreased (Investigations) | 1 (4)
Platelet count decreased (Investigations) | 1 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination lead to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes